CLINICAL TRIAL: NCT03016897
Title: ALS Testing Through Home-based Outcome Measures (ALS AT HOME)
Brief Title: ALS Testing Through Home-based Outcome Measures
Acronym: ALS AT HOME
Status: Completed | Type: Observational
Sponsor: Jeremy Shefner (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jeremy Shefner, Senior Vice President, Barrow Neurological Institute
Organization: Barrow Neurological Institute (Other)
Other Study IDs: BNI_ALS_001
Record Dates: First submitted 2016-12-22; First posted 2017-01-11 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; neurodegenerative
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Participants enrolled solely in ALS AT HOME Outcome measurement devices will be provided. Respirometer, Handgrip Meter, Skulpt Chisel, ActigraphyMeter
  Interventions: Other: Respirometer, Handgrip Meter, Skulpt Chisel, ActigraphyMeter
- Group 2: Current participants of the Answer ALS study Outcome measurement devices will be provided. Respirometer, Handgrip Meter, Skulpt Chisel, ActigraphyMeter
  Interventions: Other: Respirometer, Handgrip Meter, Skulpt Chisel, ActigraphyMeter
- Group 3: Participants without neurological disease (controls) Outcome measurement devices will be provided. Respirometer, Handgrip Meter, Skulpt Chisel, ActigraphyMeter
  Interventions: Other: Respirometer, Handgrip Meter, Skulpt Chisel, ActigraphyMeter

INTERVENTIONS:
Other: Respirometer, Handgrip Meter, Skulpt Chisel, ActigraphyMeter — Respirometer, Handgrip Meter, Skulpt Chisel, ActigraphyMeter

SUMMARY:
ALS AT HOME is a single-center study of up to 150 participants being done to determine the extent to which frequent sampling can improve the qualities of outcome measures collected at home by study participants.

DETAILED DESCRIPTION:
ALS AT HOME is a single-center study of up to 150 participants being done to determine the extent to which frequent sampling can improve the qualities of outcome measures collected at home by study participants.

The objectives of this study are to

1. assess the extent to which frequent sampling can reduce variability for the following outcome measures in ALS patients: ALSFRS-R, quantitative hand grip, pulmonary function, EIM in 4 extremities, and actigraphy and voice/speech tracking;
2. assess the compliance of ALS patients in obtained outcome measures at home over the course of 9 months;
3. directly compare outcome measures collected by patients with measurements obtained at study sites at less frequent intervals by co-enrolling 50 patients participating in the Answer ALS study; and
4. provide information to Answer ALS to more fully characterize patients in that study.

The study proposed here will assess the extent to which reducing variability of measurement through frequent sampling can reduce both sample size and duration of clinical trials, provide a first-of-its-kind detailed assessment of disease progression, and evaluate an entirely new paradigm for patient participation in such trials without the need to be geographically yoked to a clinical study center. An important component of this proposal is to jointly recruit 50 patients who also participate in the Answer ALS study that intends to generate 1000 IP cell lines from patients who receive ongoing assessment at 5 clinical sites. The 100 participants that will be co-enrolled in Answer ALS and ALS AT HOME will perform outcome measures at home in addition to having outcome measures performed at clinic sites through Answer ALS participation. Therefore, the investigators will be able to directly assess how the measures obtained by patients at home relate to those obtained by a trained evaluator at a study center using standard metrics. The investigators will also provide all data generated at home to the Answer ALS investigators, further increasing the phenotypic data available for that project.

ELIGIBILITY:
Inclusion Criteria:

* male or female, age 18 to 85 years old,
* ownership of a Smart Device (phone, tablet, etc) with Bluetooth capabilities,
* continuous internet access at home,
* willing and able to provide informed consent in compliance with the regulatory requirements through a web based interface,
* definite, Probable, or Possible ALS by modified El Escorial criteria, as documented by medical records, with duration from diagnosis 60 months or less, and
* for the 50 participants in Group 2, participation in the Answer ALS study.

Exclusion Criteria:

* diagnosed and actively undergoing treatment for cancer, heart failure, end stage renal disease, or another significant medical condition deemed by the PI to likely affect the participant's ability to comply with the protocol,
* unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the participant's ability to comply with the protocol,
* any other reasons that, in the opinion of the PI, the candidate is determined to be unsuitable for entry into the study.
* Healthy volunteers who have family members with ALS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS patient volunteers will be invited to participate in this study as well as healthy subjects for the control group.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Function | Daily for the first 3 months; for the subsequent 6 months measures will be obtained twice weekly
  Respirometer
Change in Quantitative Hand Grip | Daily for the first 3 months; for the subsequent 6 months measures will be obtained twice weekly
  Digital Handgrip Meter
Change in Electrical Impedance Myography (EIM) Measurements | Daily for the first 3 months; for the subsequent 6 months measures will be obtained twice weekly
  Skulpt Chisel
Change in Actigraphy | Daily for the first 3 months; for the subsequent 6 months measures will be obtained twice weekly
  Activity Band
ALSFRS-R | Weekly up to 9 months
  Questionnaire
Change in Patient-reported Experience measures (PREMs) | At Week 1, and then at 3, 6, and 9 months
  Questionnaire
Adverse Events | Monthly up to 9 months
  Questionnaire
Change in Voice/Speech Tracking | Daily for the first 3 months; for the subsequent 6 months measures will be obtained twice weekly
  Smartphone application

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Shefner, MD, Principal Investigator — Barrow Neurological Institute
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared with researchers conducting the Answer ALS study. It will be available through the GUID.